CLINICAL TRIAL: NCT01077596
Title: Post-marketing Carcinogenicity Study of Bupropion
Brief Title: Carcinogenicity Study of Bupropion
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111982; EPI40463; WEUKSTV1113
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Results first posted 2011-02-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Depressive Disorder; Cancer
Keywords: Carcinogenicity; Case control; Bupropion
MeSH Terms: conditions — Depressive Disorder; Neoplasms | interventions — Selective Serotonin Reuptake Inhibitors; Antidepressive Agents, Tricyclic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- New users of antidepressants Jan. 1, 1996 to Dec. 31, 2006: All new users of antidepressants January 1, 1996 through December 31, 2006. Individuals 18 years of age or older with medical and pharmacy benefits and at least 6 months of health plan enrollment before the first antidepressant prescription.
  Interventions: Drug: Regular bupropion use; Drug: Regular SSRI (Selective serotonin reuptake inhibitors) use; Drug: Regular TCA (Tricyclic antidepressants) use; Drug: Regular use of any other antidepressant

INTERVENTIONS:
Drug: Regular bupropion use — Regular use of bupropion is defined as use at least 4 times per week for at least 3 continuous months at least 12 months before index date.
Drug: Regular SSRI (Selective serotonin reuptake inhibitors) use — Regular use of SSRI is defined as use at least 4 times per week for at least 3 continuous months at least 12 months before index date.
Drug: Regular TCA (Tricyclic antidepressants) use — Regular use of TCA is defined as use at least 4 times per week for at least 3 continuous months at least 12 months before index date.
Drug: Regular use of any other antidepressant — Regular use of any other antidepressants is defined as use at least 4 times per week for at least 3 continuous months at least 12 months before index date. An "other antidepressant" would be any antidepressant other than bupropion, a SSRI or a TCA.

SUMMARY:
There is a lack of toxicology data on one bupropion metabolite, and limited literature examining bupropion use and cancer risk. This study evaluates the association between bupropion exposure and the development of cancer of the prostate, breast, lung, colon/rectum, urinary bladder, and uterus by comparing the risk of cancer in bupropion users with other antidepressant users. Because there is no evidence that bupropion is associated with any particular cancer, we have chosen the six most common cancers diagnosed in the United States to optimize statistical power/precision for cancer-site specific comparisons. Two US population-based data resources with automated claims, pharmacy, and tumor registry data are included in this study. Using a nested case-control design, this study will compare the incidence of cancer in patients exposed to bupropion with the incidence in patients exposed to other antidepressants.

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Cancers diagnosed within 12 months of initiation (i.e., new use) of antidepressant pharmacotherapy will be excluded to account for a minimum period for the development of cancer (cancer latency) and to be consistent with other studies of antidepressants and cancer.
* Patients with a history of any cancer (cancer diagnosis recorded in the tumor registries anytime before the first antidepressant prescription recorded during the study period)
* Any antidepressant use within 6 months of January 1, 1996

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New users of antidepressants January 1, 1996 through December 31, 2006, regardless of indication for use (depression, smoking cessation, other) in Henry Ford Health System and Kaiser Permanente Health Plan of Northern California. The study population is limited to individuals 18 years of age or older with medical and pharmacy benefits and at least 6 months of health plan enrollment before the first antidepressant prescription. Patients with a history of any cancer (cancer diagnosis recorded in the tumor registries anytime before the first antidepressant prescription recorded during the study period) are excluded. Cases and controls will be selected from this cohort of antidepressant-exposed study subjects.
Sampling Method: Non-Probability Sample
Enrollment: 50430 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.
Groups:
- New Antidepressant Exposure in Colorectal Cancer: Cases: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Colorectal Cancer: Cases
- New Antidepressant Exposure in Colorectal Cancer: Controls: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Colorectal Cancer: Controls
- New Antidepressant Exposure in Lung Cancer: Cases: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Lung Cancer: Cases
- New Antidepressant Exposure in Lung Cancer: Controls: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Lung Cancer: Controls
- New Antidepressant Exposure in Bladder Cancer: Cases: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Bladder Cancer: Cases
- New Antidepressant Exposure in Bladder Cancer: Controls: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Bladder Cancer: Controls
- Antidepressant Exposure in Uterine Cancer: Cases: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Uterine Cancer: Cases
- New Antidepressant Exposure in Uterine Cancer: Controls: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Uterine Cancer: Controls
- New Antidepressant Exposure in Breast Cancer: Cases: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Breast Cancer: Cases
- New Antidepressant Exposure in Breast Cancer: Controls: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Breast Cancer: Controls
- New Antidepressant Exposure in Prostate Cancer: Cases: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Prostate Cancer: Cases
- New Antidepressant Exposure in Prostate Cancer: Controls: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Prostate Cancer: Controls
Period: Overall Study
Arm/Group | New Antidepressant Exposure in Colorectal Cancer: Cases | New Antidepressant Exposure in Colorectal Cancer: Controls | New Antidepressant Exposure in Lung Cancer: Cases | New Antidepressant Exposure in Lung Cancer: Controls | New Antidepressant Exposure in Bladder Cancer: Cases | New Antidepressant Exposure in Bladder Cancer: Controls | Antidepressant Exposure in Uterine Cancer: Cases | New Antidepressant Exposure in Uterine Cancer: Controls | New Antidepressant Exposure in Breast Cancer: Cases | New Antidepressant Exposure in Breast Cancer: Controls | New Antidepressant Exposure in Prostate Cancer: Cases | New Antidepressant Exposure in Prostate Cancer: Controls
Started | 350 | 1050 | 457 | 1370 | 294 | 882 | 308 | 837 | 2842 | 28420 | 2215 | 22150
Completed | 350 | 1050 | 457 | 1370 | 294 | 882 | 308 | 837 | 2842 | 28420 | 2215 | 22150
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- New Antidepressant Exposure in Uterine Cancer: Cases: New Antidepressant Exposure (defined as no antidepressant exposure within previous 6 months) in Uterine Cancer: Cases
- Total: Total of all reporting groups
Arm/Group | New Antidepressant Exposure in Colorectal Cancer: Cases | New Antidepressant Exposure in Colorectal Cancer: Controls | New Antidepressant Exposure in Lung Cancer: Cases | New Antidepressant Exposure in Lung Cancer: Controls | New Antidepressant Exposure in Bladder Cancer: Cases | New Antidepressant Exposure in Bladder Cancer: Controls | New Antidepressant Exposure in Uterine Cancer: Cases | New Antidepressant Exposure in Uterine Cancer: Controls | New Antidepressant Exposure in Breast Cancer: Cases | New Antidepressant Exposure in Breast Cancer: Controls | New Antidepressant Exposure in Prostate Cancer: Cases | New Antidepressant Exposure in Prostate Cancer: Controls | Total
Number analyzed (Participants) | 350 | 1050 | 457 | 1370 | 294 | 882 | 308 | 837 | 2842 | 28420 | 2215 | 22150 | 61175
Age, Customized [Number; unit: Participants]
  45-54 years | 34 | 102 | 47 | 140 | 17 | 51 | 59 | 172 | 678 | 6780 | 193 | 1930 | 10203
  55-64 years | 73 | 219 | 102 | 306 | 63 | 189 | 90 | 245 | 849 | 8490 | 669 | 6690 | 17985
  65-74 years | 119 | 357 | 159 | 477 | 104 | 312 | 84 | 224 | 707 | 7070 | 877 | 8770 | 19260
  >=75 years | 124 | 372 | 149 | 447 | 110 | 330 | 75 | 196 | 608 | 6080 | 476 | 4760 | 13727
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 378 | 175 | 525 | 91 | 273 | 308 | 837 | 2842 | 28420 | 0 | 0 | 33975
  Male | 224 | 672 | 282 | 845 | 203 | 609 | 0 | 0 | 0 | 0 | 2215 | 22150 | 27200
Number of participants diagnosed with the indicated conditions and using the indicated therapies [Number; unit: participants] — A value of "0" indicates that no data are available for that particular treatment arm. Smoking status data were not collected for breast cancer and prostate cancer cases and controls, as it is not a necessary variable for analysis. NSAIDS, non-steroidal anti-inflammatory drugs.
  participants
    Exposed to multiple antidepressants | 47 | 160 | 62 | 191 | 44 | 147 | 53 | 162 | 564 | 5756 | 340 | 3782 | 11308
    Ever smokers | 252 | 643 | 428 | 772 | 247 | 573 | 142 | 389 | 0 | 0 | 0 | 0 | 3446
    Unknown smoking status | 4 | 70 | 5 | 183 | 1 | 29 | 4 | 27 | 0 | 0 | 0 | 0 | 323
    Ever diagnosed (dx) with depression | 110 | 329 | 108 | 408 | 83 | 273 | 119 | 319 | 1091 | 10541 | 677 | 6700 | 20758
    Ever dx with inflammatory bowel disease (IBD) | 1 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
    Users of oral contraceptives (OC) | 6 | 7 | 0 | 0 | 0 | 0 | 8 | 45 | 236 | 1987 | 0 | 0 | 2289
    Users of hormone replacement therapy (HRT) | 57 | 225 | 0 | 0 | 0 | 0 | 153 | 441 | 1796 | 17184 | 0 | 0 | 19856
    Users of NSAIDs | 269 | 859 | 370 | 1123 | 0 | 0 | 0 | 0 | 2340 | 23730 | 1800 | 17887 | 48378

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Diagnosed With Any of the Cancers Under Investigation Who Were Regularly Exposed to the Indicated Antidepressant
Description: The following are the cancers under investigation: colorectal, lung, bladder, uterus, breast, and prostate. Cancer case were nested within a cohort of new antidepressant users. New antidepressant users were defined as no previous antidepressant prescription in the previous 6 months. Cases were identified and matched with controls from the same new-user cohort. Cal year, calendar year; dx, diagnosis; IBD, Inflammatory Bowel Disease; OC, oral contraceptive; HRT/ERT, hormone replacement therapy/estrogen replacement therapy; NSAID, non-steroidal anti-inflammatory drug.
Time Frame: January 1, 1996 - December 31, 2006
Population: Participants diagnosed with colorectal, lung, bladder, uterus, breast, or prostate cancer who were new antidepressant users
Measure: Number; unit: participants
Groups:
- Bupropion, Regular Use: Regular Bupropion use was defined as 4 times per week for 3 months at least 12 months before index date
- All Non-bupropion Antidepressants, Regular Use: Regular antidepressant use of non-bupropion was defined as use of non-bupropion antidepressant for 4 times per week for 3 months at least 12 months before index date
- Tricyclic Antidepressants (TCA), Regular Use: Regular TCA use was defined as use of TCA for 4 times per week for 3 months at least 12 months before index date
- Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use: Regular SSRI use was defined as use of SSRI antidepressant for 4 times per week for 3 months at least 12 months before index date
- Other Antidepressants, Regular Use: Regular "other" antidepressant use was defined as use other antidepressant aside from Bupropion, TCA, and SSRI for 4 times per week for 3 months at least 12 months before index date
Arm/Group | Bupropion, Regular Use | All Non-bupropion Antidepressants, Regular Use | Tricyclic Antidepressants (TCA), Regular Use | Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use | Other Antidepressants, Regular Use
Number analyzed (Participants) | 8038 | 42392 | 18537 | 23740 | 10123
participants
  Cases | 853 | 4561 | 1963 | 2570 | 1027
  Controls | 6332 | 37831 | 16574 | 21170 | 9096
Statistical Analysis 1: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.2, 95% CI [1.1 to 1.3]
Statistical Analysis 2: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.1, 95% CI [1.0 to 1.2] — Adjusted for age, sex, cal year, study site, tumor characteristics, multiple antidepressants exposure, smoking, hysterectomy status, previous depression dx, previous IBD diagnosis, OC use, HRT/ERT use, and NSAID use
Statistical Analysis 3: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.2, 95% CI [1.1 to 1.3]
Statistical Analysis 4: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.1, 95% CI [1.0 to 1.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.2, 95% CI [1.0 to 1.3]
Statistical Analysis 6: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.1, 95% CI [1.0 to 1.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.2, 95% CI [1.1 to 1.4]
Statistical Analysis 8: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.2, 95% CI [1.0 to 1.3] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Number of Participants Diagnosed With Colorectal Cancer Who Were Regularly Exposed to the Indicated Antidepressant
Description: In this outcome, colorectal cancer is under investigation: Cancer case were nested within a cohort of new antidepressant users. New antidepressant users were defined as no previous antidepressant prescription in the previous 6 months. Colorectal cancer cases were identified and matched with controls from the same new-user cohort. Cal year, calendar year; dx, diagnosis; IBD, Inflammatory Bowel Disease; OC, oral contraceptive; HRT/ERT, hormone replacement therapy/estrogen replacement therapy; NSAID, non-steroidal anti-inflammatory drug.
Time Frame: January 1, 1996 - December 31, 2006
Population: Participants diagnosed with colorectal cancer who were new antidepressant users.
Measure: Number; unit: participants
Groups:
- Tricyclic Antidepressants (TCA), Regular Use: Regular TCA use was defined as use of tricyclic antidepressant for 4 times per week for 3 months at least 12 months before index date
- Other Antidepressants, Regular Use: Regular 'other' antidepressant use was defined as use other antidepressant aside from Bupropion, TCA and SSRI for 4 times per week for 3 months at least 12 months before index date
Arm/Group | Bupropion, Regular Use | All Non-bupropion Antidepressants, Regular Use | Tricyclic Antidepressants (TCA), Regular Use | Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use | Other Antidepressants, Regular Use
Number analyzed (Participants) | 126 | 973 | 432 | 545 | 201
participants
  Cases | 37 | 234 | 111 | 134 | 35
  Controls | 89 | 739 | 321 | 411 | 166
Statistical Analysis 1: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.4, 95% CI [0.9 to 2.2]
Statistical Analysis 2: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.2, 95% CI [0.8 to 2.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.2, 95% CI [0.8 to 2.0]
Statistical Analysis 4: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.1, 95% CI [0.7 to 1.9] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.3, 95% CI [0.8 to 2.1]
Statistical Analysis 6: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.1, 95% CI [0.7 to 1.9] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 2.2, 95% CI [1.2 to 3.9]
Statistical Analysis 8: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 2.0, 95% CI [1.1 to 3.6] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Number of Participants Diagnosed With Lung Cancer Who Were Regularly Exposed to the Indicated Antidepressant
Description: In this outcome, lung cancer is under investigation: Cancer case were nested within a cohort of new antidepressant users. New antidepressant users were defined as no previous antidepressant prescription in the previous 6 months. Lung cancer cases were identified and matched with controls from the same new-user cohort. Cal year, calendar year; dx, diagnosis; IBD, Inflammatory Bowel Disease; OC, oral contraceptive; HRT/ERT, hormone replacement therapy/estrogen replacement therapy; NSAID, non-steroidal anti-inflammatory drug.
Time Frame: January 1, 1996 - December 31, 2006
Population: Participants diagnosed with lung cancer who were new antidepressant users.
Measure: Number; unit: participants
Arm/Group | Bupropion, Regular Use | All Non-bupropion Antidepressants, Regular Use | Tricyclic Antidepressants (TCA), Regular Use | Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use | Other Antidepressants, Regular Use
Number analyzed (Participants) | 240 | 1172 | 498 | 670 | 233
participants
  Cases | 115 | 250 | 109 | 138 | 47
  Controls | 125 | 922 | 389 | 532 | 186
Statistical Analysis 1: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 4.5, 95% CI [3.2 to 6.3]
Statistical Analysis 2: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 3.0, 95% CI [2.0 to 4.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 4.0, 95% CI [2.8 to 5.8]
Statistical Analysis 4: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 2.9, 95% CI [1.9 to 4.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 4.4, 95% CI [3.1 to 6.3]
Statistical Analysis 6: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 3.0, 95% CI [1.9 to 4.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 4.5, 95% CI [2.8 to 7.2]
Statistical Analysis 8: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 3.5, 95% CI [2.1 to 5.9] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Number of Participants Diagnosed With Bladder Cancer Who Were Regularly Exposed to the Indicated Antidepressant
Description: In this outcome, bladder cancer is under investigation: Cancer case were nested within a cohort of new antidepressant users. New antidepressant users were defined as no previous antidepressant prescription in the previous 6 months. Bladder cancer cases were identified and matched with controls from the same new-user cohort. Cal year, calendar year; dx, diagnosis; IBD, Inflammatory Bowel Disease; OC, oral contraceptive; HRT/ERT, hormone replacement therapy/estrogen replacement therapy; NSAID, non-steroidal anti-inflammatory drug.
Time Frame: January 1, 1996 - December 31, 2006
Population: Participants diagnosed with bladder cancer who were new antidepressant users.
Measure: Number; unit: participants
Arm/Group | Bupropion, Regular Use | All Non-bupropion Antidepressants, Regular Use | Tricyclic Antidepressants (TCA), Regular Use | Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use | Other Antidepressants, Regular Use
Number analyzed (Participants) | 125 | 853 | 385 | 454 | 199
participants
  Cases | 48 | 191 | 88 | 103 | 40
  Controls | 77 | 662 | 297 | 351 | 159
Statistical Analysis 1: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 2.6, 95% CI [1.7 to 4.1]
Statistical Analysis 2: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 2.1, 95% CI [1.3 to 3.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 2.3, 95% CI [1.4 to 3.6]
Statistical Analysis 4: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.8, 95% CI [1.1 to 3.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 2.3, 95% CI [1.5 to 3.7]
Statistical Analysis 6: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.8, 95% CI [1.1 to 3.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 2.6, 95% CI [1.5 to 4.5]
Statistical Analysis 8: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 2.2, 95% CI [1.3 to 3.9] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Number of Participants Diagnosed With Uterine Cancer Who Were Regularly Exposed to the Indicated Antidepressant
Description: In this outcome, uterine cancer is under investigation: Cancer case were nested within a cohort of new antidepressant users. New antidepressant users were defined as no previous antidepressant prescription in the previous 6 months. Uterine cancer cases were identified and matched with controls from the same new-user cohort. Cal year, calendar year; dx, diagnosis; IBD, Inflammatory Bowel Disease; OC, oral contraceptive; HRT/ERT, hormone replacement therapy/estrogen replacement therapy; NSAID, non-steroidal anti-inflammatory drug.
Time Frame: January 1, 1996 - December 31, 2006
Population: Participants diagnosed with uterine cancer who were new antidepressant users.
Measure: Number; unit: participants
Arm/Group | Bupropion, Regular Use | All Non-bupropion Antidepressants, Regular Use | Tricyclic Antidepressants (TCA), Regular Use | Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use | Other Antidepressants, Regular Use
Number analyzed (Participants) | 116 | 866 | 371 | 484 | 210
participants
  Cases | 25 | 233 | 114 | 124 | 45
  Controls | 91 | 633 | 257 | 360 | 165
Statistical Analysis 1: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 0.8, 95% CI [0.5 to 1.3]
Statistical Analysis 2: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 0.7, 95% CI [0.4 to 1.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 0.6, 95% CI [0.4 to 1.1]
Statistical Analysis 4: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 0.6, 95% CI [0.3 to 1.0] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 0.8, 95% CI [0.5 to 1.4]
Statistical Analysis 6: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 0.8, 95% CI [0.4 to 1.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.1, 95% CI [0.6 to 2.0]
Statistical Analysis 8: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.0, 95% CI [0.6 to 1.9] — Adjusted for age, sex, cal year, study site, tumor characteristics, multiple antidepressants exposure, smoking, hysterectomy status†, previous depression dx, previous IBD‡ diagnosis, OC§ use, HRT/ERT use, and NSAID use

6. Secondary Outcome: Number of Participants Diagnosed With Breast Cancer Who Were Regularly Exposed to the Indicated Antidepressant
Description: In this outcome, breast cancer is under investigation: Cancer case were nested within a cohort of new antidepressant users. New antidepressant users were defined as no previous antidepressant prescription in the previous 6 months. Breast cancer cases were identified and matched with controls from the same new-user cohort. Cal year, calendar year; dx, diagnosis; IBD, Inflammatory Bowel Disease; OC, oral contraceptive; HRT/ERT, hormone replacement therapy/estrogen replacement therapy; NSAID, non-steroidal anti-inflammatory drug.
Time Frame: January 1, 1996 - December 31, 2006
Population: Participants diagnosed with breast cancer who were new antidepressant users.
Measure: Number; unit: participants
Arm/Group | Bupropion, Regular Use | All Non-bupropion Antidepressants, Regular Use | Tricyclic Antidepressants (TCA), Regular Use | Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use | Other Antidepressants, Regular Use
Number analyzed (Participants) | 3268 | 23361 | 10279 | 13454 | 5638
participants
  Cases | 302 | 2173 | 941 | 1265 | 497
  Controls | 2966 | 21188 | 9338 | 12189 | 5141
Statistical Analysis 1: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 0.9, 95% CI [0.8 to 1.1]
Statistical Analysis 2: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 0.9, 95% CI [0.8 to 1.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.0, 95% CI [0.9 to 1.2]
Statistical Analysis 4: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.0, 95% CI [0.8 to 1.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.0, 95% CI [0.8 to 1.1]
Statistical Analysis 6: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 0.9, 95% CI [0.8 to 1.1] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.1, 95% CI [0.9 to 1.3]
Statistical Analysis 8: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.1, 95% CI [0.9 to 1.2] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Number of Participants Diagnosed With Prostate Cancer Who Were Regularly Exposed to the Indicated Antidepressant
Description: In this outcome, prostate cancer is under investigation: Cancer case were nested within a cohort of new antidepressant users. New antidepressant users were defined as no previous antidepressant prescription in the previous 6 months. Prostate cancer cases were identified and matched with controls from the same new-user cohort. Cal year, calendar year; dx, diagnosis; IBD, Inflammatory Bowel Disease; OC, oral contraceptive; HRT/ERT, hormone replacement therapy/estrogen replacement therapy; NSAID, non-steroidal anti-inflammatory drug.
Time Frame: January 1, 1996 - December 31, 2006
Population: Participants diagnosed with prostate cancer who were new antidepressant users.
Measure: Number; unit: participants
Arm/Group | Bupropion, Regular Use | All Non-bupropion Antidepressants, Regular Use | Tricyclic Antidepressants (TCA), Regular Use | Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use | Other Antidepressants, Regular Use
Number analyzed (Participants) | 3550 | 17042 | 7436 | 9112 | 4089
participants
  Cases | 326 | 1480 | 600 | 806 | 363
  Controls | 3224 | 15562 | 6836 | 8306 | 3726
Statistical Analysis 1: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.1, 95% CI [1.0 to 1.3]
Statistical Analysis 2: Comparison: Bupropion, Regular Use vs All Non-bupropion Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.2, 95% CI [1.0 to 1.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.2, 95% CI [1.0 to 1.4]
Statistical Analysis 4: Comparison: Bupropion, Regular Use vs Tricyclic Antidepressants (TCA), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.2, 95% CI [1.0 to 1.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.1, 95% CI [0.9 to 1.2]
Statistical Analysis 6: Comparison: Bupropion, Regular Use vs Selective Serotonin Reuptake Inhibitors (SSRI), Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.1, 95% CI [0.9 to 1.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Crude Odds Ratio = 1.0, 95% CI [0.9 to 1.2]
Statistical Analysis 8: Comparison: Bupropion, Regular Use vs Other Antidepressants, Regular Use; Test type: Superiority or Other; Adjusted Odds Ratio = 1.0, 95% CI [0.8 to 1.2] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing data; thus, no assessments for Serious or Non-serious Adverse Events were performed.
Arm/Group | New Antidepressant Exposure in Colorectal Cancer: Cases | New Antidepressant Exposure in Colorectal Cancer: Controls | New Antidepressant Exposure in Lung Cancer: Cases | New Antidepressant Exposure in Lung Cancer: Controls | New Antidepressant Exposure in Bladder Cancer: Cases | New Antidepressant Exposure in Bladder Cancer: Controls | New Antidepressant Exposure in Uterine Cancer: Cases | New Antidepressant Exposure in Uterine Cancer: Controls | New Antidepressant Exposure in Breast Cancer: Cases | New Antidepressant Exposure in Breast Cancer: Controls | New Antidepressant Exposure in Prostate Cancer: Cases | New Antidepressant Exposure in Prostate Cancer: Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.